CLINICAL TRIAL: NCT03716947
Title: A Randomized Controlled Study Between Mechanical and a Viscoelastic Disc Prosthesis in the Lumbar Spine. A Comparison on Clinical Outcome and Facet-joint Load Between Two Different TDR Designs.
Brief Title: A Comparative Study Between Mechanical and a Viscoelastic Disc Prosthesis in the Lumbar Spine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Svante Berg, MD, PhD, Associate Professor, Senior Consultant, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: mojje
Record Dates: First submitted 2018-07-12; First posted 2018-10-23 (Actual); Last update posted 2020-12-16 (Actual); Status verified 2020-12

CONDITIONS: Degenerative Disc Disease; Discogenic Low Back Pain
Keywords: Clinical outcome; Mobility; Facet-joints
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ORBIT Mechanical disc prosthesis (Active Comparator): Surgical procedure with total disc replacement using mechanical disc prosthesis device, "ORBIT, Globus Medical"
  Interventions: Procedure: Device: ZACK
- ZACK viscoelastic disc prosthesis (Experimental): Surgical procedure with total disc replacement using viscoelastic disc prosthesis device, "ZACK, FH Orthopaedics"
  Interventions: Procedure: Device: ORBIT
- ORBIT SASCA (Active Comparator): Surgical procedure with total disc replacement (TDR) using ORBIT disc prostheses device combined with adjacent level anterior intracorporal fusion (ALIF) with intracorporal device SASCA.
  Interventions: Procedure: Device: ZACK; Procedure: Device: SASCA
- ZACK SASCA (Experimental): Surgical procedure with total disc replacement (TDR) using ZACK disc prostheses device combined with adjacent level anterior intracorporal fusion (ALIF) with intracorporal device SASCA.
  Interventions: Procedure: Device: ORBIT; Procedure: Device: SASCA

INTERVENTIONS:
Procedure: Device: ZACK — Surgical procedure with total disc replacement using ZACK disc prostheses
  Arms: ORBIT Mechanical disc prosthesis; ORBIT SASCA
Procedure: Device: ORBIT — Surgical procedure with total disc replacement using ORBIT disc prostheses
  Arms: ZACK SASCA; ZACK viscoelastic disc prosthesis
Procedure: Device: SASCA — Surgical procedure with anterior intracorporal fusion (ALIF) combined with adjacent level total disc replacement (TDR) (using either ORBIT mechanical disc prosthesis or ZACK viscoelastic disc prosthesis)
  Arms: ORBIT SASCA; ZACK SASCA

SUMMARY:
TDR implants for the lumbar spine are currently most 2- or 3-piece devices with a purely mechanical function that provide/restore mobility. Lately interest is growing on non-mechanical implants that could possibly provide/restore mobility, but also produce counterforces on mobility as in healthy discs. No previous comparison between these two concepts has been performed, neither on clinical outcome, neither on specific differences on facet-joint load and wear.

DETAILED DESCRIPTION:
A total of 250 patients are to be enrolled and treated. Inclusion criteria is unbearable pain and dysfunction from degenerative disc disease (DDD) that at one or two segments in the lover lumbar spine, that has not responded positively from at least one year of conservative treatment (that is combination of intense physical training and drugs).

Patients with DDD below L3 vertebra are divided I three groups:

1. One segment DDD appropriate for treatment with TDR.
2. Two segments DDD appropriate for treatment with TDR.
3. One segment DDD appropriate for treatment with TDR and one segment DDD not appropriate for treatment with TDR, that will be treated with anterior fusion (ALIF) at the same surgical procedure, called "hybrids". Within all three groups there will be an equal randomization between the two prosthesis types.

Clinical outcome will be evaluated from questionnaires sent out to patients after 12- and 24 months and 5- and 10 years after surgery. The questionnaire are the currently used ones from the Swedish Spine Registry (SweSpine) including VAS leg/back, EuroQol ,GA and ODI. Complications will be registered continuously and facet-joint load/health will be examined from flex-ext x-rays at 1 and 2 years. At the 2-year check up a 3D-CT will be performed to further evaluate the facet joints and their load under flex-ext.

ELIGIBILITY:
Inclusion Criteria:

* Incapacitating pain from DDD (both clinical and radiological) in one or two segments below the L3 vertebra, were at least one segment is suitable for TDR treatment.
* Patient with more than one year of pain, that has during this period made a prolonged and adequate conservative program.

-Patient between 20 and 55 years of age. -

-Patient able to understand written and spoken Swedish.

Exclusion Criteria:

* Patient does not accept to be part of the study.
* Three or more segments suspected to be symptomatic.
* Earlier vertebral fracture, tumour, infection or fusion in the lumbar spine. -Substantial scoliosis/deformity.
* Need for posterior decompression.
* Pregnancy, psychiatric illness or drug abuse. -Patient does not understand written and spoken Swedish and can thus not take part in information and answer questionnaires.

-Patient residing outside Sweden and thus is not covered with SweSpine. -

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 246 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Patient reported back pain after two years in Swespine national registry | 2, 5, 10 years
  GA (Global Assessment of back pain, patient-based evaluation of leg and back pain as compared to preoperatively,1-5, 1 disappeared and 5 worsened) ,collected from questionnaires

SECONDARY OUTCOMES:
VAS, Visual Analogue Scale | 2, 5, 10 years
  VAS (Visual Analogue Scale, 0 no pain, 100 worst possible pain) of back and leg,collected from questionnaires
ODI, Oswestry disability index | 2, 5, 10 years
  ODI (Oswestry disability index, self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel, 0-5 zero indicating the least amount of disability and 5 indicating most severe disability)
EQ-5D, Health-related quality of life | 2, 5, 10 years
  EuroQol EQ-5D-5L, Self-completed questionnaire regarding mobility, self-care, usual activities, pain/discomfort and anxiety/depression. EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Re-operation related to facet-joint arthritis | 2, 5, 10 years
  Medical records, questionnaires and further registrations in SweSpine reporting repeat surgery, with a differentiation of the medical reason for that intervention.
Facet-joint pathology prevalence | 2, 5, 10 years
  Prevalence of radiological signs of arthritis or ankylosis from flex-ext X-rays and 3D-CT
Postoperative complications | Two years after the last patient is treated
  Medical records will be evaluated for surgically related complications, death, infection, bleeding, implant loosening, re-operation/revision, neurological complication, thrombosis, implant failure, implant malpositioning/displacement, non-union, incisional hernia, retrograde ejaculation

CONTACTS AND LOCATIONS:
Overall Officials: Svante Berg, MD,PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Stockholm Spine Center, Stockholm, Upplands Väsby, Sweden

IPD SHARING:
Plan to Share IPD: No